CLINICAL TRIAL: NCT00861484
Title: A Double Blind, Parallel Group, Placebo Controlled Study to Evaluate the Effect of a Single Oral Dose of GSK958108 on Ejaculatory Latency Time (ELT) in Male Patient Suffering From Premature Ejaculation
Brief Title: Proof of Mechanism in ELT
Acronym: PoM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111155
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK958108 3 mg (Experimental): Experimental
  Interventions: Drug: GSK958108
- Placebo of GSK958108 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK958108 — Coated Tablets 1 mg
  Arms: GSK958108 3 mg
Drug: Placebo — Coated tablets
  Arms: Placebo of GSK958108

SUMMARY:
The purpose of this study is to determine if the administration of GSK958108 can delay ejaculation in patients with primary premature ejaculation as measured by the ejaculatory latency time (ELT) using the masturbation model and sexual visual stimulation, and to evaluate the safety and tolerability of GSK958108 in healthy men with PE

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual male subject with self-reported moderate or severe primary Premature ejaculation with ejaculation occurring on or before penetration, or shortly there after with minimal stimulation
* Baseline Ejaculation Latency time < 3 minutes
* Subjects must agree to use a contraception methods as per protocol
* Body weight > or = 50 kg and Body Mass Index within the range 19.0-29.9 Kg/m2
* Subject with normal visual acuity (with appropriate correction if needed)
* Subject able to cooperate in all study procedure including the eye examination with use of mydriatics

Exclusion Criteria:

* Erectile dysfunction
* History of migraine
* Current clinically relevant abnormality
* History of psychiatric illness or suicidal attempts or behaviours
* History of any eye disorder or colour blind, excluding myopia and presbyopia
* Cardiac conduction disorder or other clinically significant cardiac disease
* Positive at pre-study drug/alcohol screen and to Hepatitis or HIV tests
* Regular consumption of alcohol
* History of sensitivity or intolerance to drugs
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice [and/or pummelos, exotic citrus fruits, grapefruit hybrids] from 7 days prior to the first dose of study medication
* Subject has received or is continuing to receive any treatment for premature ejaculation in the four weeks prior to the study start
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements prior to the first dose of study medication
* Participation in another clinical trial in the previous month
* Exposure to more than four new experimental drugs within the previous 12 months
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2008-11-26 (Actual); Primary Completion 2009-12-11 (Actual); Study Completion 2009-12-11 (Actual)

PRIMARY OUTCOMES:
Time to achieve ejaculation from the start of masturbation during audio-video erotic stimuli | 50 minutes

SECONDARY OUTCOMES:
Safety and tolerability measured as adverse events occurrence, vital signs variations, safety laboratory, eye assessments, ECG and physical examination | 8 weeks
Blood concentration of GSK958108 at different timepoints | From predose to 30 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Verona, Veneto, Italy

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 111155 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111155?search=study&search_terms=111155#rs
- Available data/document: Study Protocol: 111155 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111155 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111155 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111155 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111155 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111155 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111155 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register